CLINICAL TRIAL: NCT06293846
Title: BeFit Toolbox Collaboration: Building Empowerment Through Fitness
Acronym: BEFIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Kimberly McCall, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-300012108; IRB Designation (Other: UAB)
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Low-Income Population; Women's Health
Keywords: Women's Health; Health Disparities; Behavior Change; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- What I Learned at Home (Experimental): What I Learned at Home is a self-efficacy behavioral intervention that will help provide the framework of implementation for the BeFIT program in the future. The BeFIT program will be a component of the WILAH framework.
  Interventions: Behavioral: What I Learned at Home

INTERVENTIONS:
Behavioral: What I Learned at Home — What I Learned at Home is a self-efficacy intervention intended to build home repair and management skills while improving performance self-efficacy.
  Other Names: WILAH

SUMMARY:
This project will identify the causative behavioral factors in low-income African American women leading to sedentarism, a major source of morbidity in HABD communities. Working with our partner, WUCN, we will engage with women in HABD housing to develop and (later) deliver a physical activity education program (BeFit) customized for this population.

DETAILED DESCRIPTION:
Despite clear evidence of improved health outcomes with regular exercise (see Bliss et al., 2021; Kleinloog et al., 20,22 for recent reviews), national statistics suggest that a mere 48% of Americans meet the recommended levels of physical activity (Centers for Disease Control and Prevention [CDC], 2018). Alarmingly, fewer than 30% of African American women living in public housing meet these recommended levels, marking the lowest rate among all demographic groups (Lee & Im, 2010; Hilland et al., 2020). Cerebrovascular disease in this population is increasing in prevalence, as is early presentation underscoring the urgent need for innovative, culturally relevant strategies to promote and study the effects of physical activity engagement within this under-resourced community (Turney et al., 2022; Zuellsdorf et al., 2020). However, developing relevant research-based interventions requires understanding and adapting specific programs to local public housing challenges (Casagrande et al., 2008). Mistrust is the primary barrier to relationship development in this population, and engagement with an established community partner is critical for local implementation. This proposal aims to develop a physical activity education program for women at high risk of disease to promote healthy lifestyles and mitigate the risk of neurological pathology.

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria for participants are as follows: female, at least 18 years of age, mothers of school-aged children (K-12), tenants of HABD in good standing with a minimum of one year of stable living arrangements, and availability during program hours.

Exclusion Criteria:

* Inability to understand study instructions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This is a women's health study investigating barriers women heads of household face in engaging in physical activity.
Enrollment: 50 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Barriers to Physical Activity Self-Report | 12 weeks
  Report of barriers to engagement in physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Kim McCall, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bliss ES, Wong RH, Howe PR, Mills DE. Benefits of exercise training on cerebrovascular and cognitive function in ageing. J Cereb Blood Flow Metab. 2021 Mar;41(3):447-470. doi: 10.1177/0271678X20957807. Epub 2020 Sep 20. PMID 32954902
- [Background] Kleinloog JPD, Nijssen KMR, Mensink RP, Joris PJ. Effects of Physical Exercise Training on Cerebral Blood Flow Measurements: A Systematic Review of Human Intervention Studies. Int J Sport Nutr Exerc Metab. 2022 Sep 27;33(1):47-59. doi: 10.1123/ijsnem.2022-0085. Print 2023 Jan 1. PMID 36170974
- [Background] Craike M, Bourke M, Hilland TA, Wiesner G, Pascoe MC, Bengoechea EG, Parker AG. Correlates of Physical Activity Among Disadvantaged Groups: A Systematic Review. Am J Prev Med. 2019 Nov;57(5):700-715. doi: 10.1016/j.amepre.2019.06.021. PMID 31630762